CLINICAL TRIAL: NCT05848908
Title: Advanced Provision of Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Alison Edelman, Clinical Instructor, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUYD00025095
Record Dates: First submitted 2023-04-28; First posted 2023-05-08 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Pregnancy Related
Keywords: Counseling, telehealth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Telehealth Visit (Experimental): telemedicine visit and follow-up surveys
  Interventions: Other: Telehealth Visit

INTERVENTIONS:
Other: Telehealth Visit — telemedicine visit and follow-up surveys

SUMMARY:
This study aims to evaluate advanced provision of an anti-progestin with a prostaglandin for future use (in the next 12 months) in individuals at risk for pregnancy but not desiring a pregnancy.

DETAILED DESCRIPTION:
The purpose of this study is to learn more about counseling via telemedicine and advanced provision of medications to individuals at risk for pregnancy but before they are pregnant. If they experience this event, then they may subsequently have immediate access to the care they need plus an established connection with a health provider.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 40 years old at time of consent
* Anatomically capable of pregnancy
* Self-reported a history of regular menses (>24 and <38 days) in the past 3 years (other than during pregnancy)
* Not currently pregnant and not desiring to be pregnant in the next year
* Say they would seek to end the pregnancy if they became pregnant in the next year and who do not express a preference for an in office procedure
* At-risk for unintended pregnancy defined as:
* those who report being sexually active (vaginal sex with partners with sperm)
* have not been told by a clinician that they cannot become pregnant
* have not had a permanent contraception procedure and whose current sexual partner(s) has not had a permanent contraception procedure
* who are not using a long-acting reversible contraceptive (LARC)
* Willing and able to provide informed consent
* Willing/able to receive phone calls from study staff and complete electronic surveys distributed by EMR or email
* Planning to live within the state of Oregon or Washington for the 12 month study period.

Exclusion Criteria:

* Less than 18 and older than 40 years old at the time of consent
* Any medical contraindications to MAB (hemorrhagic disorder or will be taking anticoagulants during study period, chronic adrenal failure or will be taking long term corticosteroids >1 week during study period, inherited porphyria, or an allergy to mifepristone or misoprostol)
* Currently pregnant or desiring pregnancy in the next year
* State they would not seek to end a pregnancy if they became pregnant in the next year or who express a preference for an in office procedure
* History of ectopic pregnancy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-06-28 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
The proportion of participants reporting confidence in key steps of taking medications | Enrollment to 12 months
  The proportion of participants reporting confidence in key steps of taking medications in follow-up surveys
Proportion of participants reporting satisfaction with the process | Enrollment to 12 months
  Proportion of participants reporting satisfaction with the process in follow up surveys

CONTACTS AND LOCATIONS:
Locations (1):
- OHSU, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No